CLINICAL TRIAL: NCT02294695
Title: Early Procalcitonin Kinetics May Indicate Effectiveness of the Empirical Antibiotic Therapy in Sepsis Within Hours
Brief Title: Early Procalcitonin Kinetics During Empirical Antibiotic Therapy in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Domonkos Trásy (Other)
Responsible Party: Sponsor-Investigator, Domonkos Trásy, Ph.D. student; Department of Anaesthesiology and Intensive Therapy, Szeged University
Organization: Szeged University (Other)
Other Study IDs: EProK study
Record Dates: First submitted 2014-11-07; First posted 2014-11-19 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2014-11

CONDITIONS: Bacterial Infections
Keywords: Empiric antibiotic therapy
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Appropriate empiric antibiotic therapy: Based on the microbiological results patients were grouped post hoc into "appropriate" and "inappropriate" groups by two independent experts (intensivist, infectologist) who were blinded for PCT.
- Inappropriate empiric antibiotic therapy: Based on the microbiological results patients were grouped post hoc into "appropriate" and "inappropriate" groups by two independent experts (intensivist, infectologist) who were blinded for PCT.

SUMMARY:
To investigate the value of procalcitonin (PCT) kinetics between 0-8-16-24 hours after starting empirical antibiotic therapy in critically ill patients, to predict appropriate or inappropriate antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of infection
* Suspected or proven acute infection requiring empiric antibiotic therapy as decided by the attending ICU physician
* Suspected site of infection has to be present and documented
* Microbiological sample sent for staining
* Inflammatory markers available at the start of the therapy

Exclusion Criteria:

* Patients younger than 18 years
* Who received prophylactic or empiric antibiotic therapy 48 hours before inclusion
* Whose receiving acute renal replacement therapy in the first 24 hours following antibiotic treatment
* Following cardiopulmonary resuscitation
* End stage diseases with a "do not resuscitate" order
* Immunocompromised patients (human immunodeficiency virus infection, bone marrow transplantation, malignant haematological disorders and chemotherapy)
* Post cardiac surgery patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years with suspected infection on admission or during their stay on the intensive care unit were screened for eligibility. Patients were enrolled, when the attending intensive care specialist had a suspicion of infection and decided to start empirical antibiotic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Procalcitonin kinetic | The first six days after starting empiric antibiotic treatment
  PCT levers are measured every 8 hours in the first day after starting empiric antibiotic treatment then daily and the changes in percentage are followed form the baseline value measured right before the first exposition of the antibiotic therapy.

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment score | The first six days after starting empiric antibiotic treatment
  SOFA score is measured every day after starting empiric antibiotic treatment.

OTHER OUTCOMES:
Length of Intensive Care Unit stay | Maximum 90 days after enrollment
Intensive Care Unit mortality | Maximum 90 days after enrollment
Length of hospital stay | Maximum 90 days after enrollment
Hospital mortality | Maximum 90 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary